CLINICAL TRIAL: NCT05533944
Title: Fast-tracking ERCP Learning: Does Training on a Mechanical Simulator Improve Trainee's Clinical Performance? A Randomized Trial To Evaluate Predictive Validity of Boškoski-Costamagna ERCP Trainer Simulator.
Brief Title: Fast-tracking ERCP Learning: Does Training on a Mechanical Simulator Improve Trainee's Clinical Performance?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Amsterdam UMC, location VUmc (Other); Universitaire Ziekenhuizen KU Leuven (Other); Hospital Nord (Other); Centre Hospitalier Universitaire de Nice (Other); Erasmus Medical Center (Other); Leiden University Medical Center (Other); The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other); Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ErasmeUH1
Record Dates: First submitted 2022-09-01; First posted 2022-09-09 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2022-09

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Simulation Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation group (Active Comparator): Trainees will undergo routine hands-on clinical ERCP training. In addition, trainees from Simulation Group have coached simulation training, by participating in three two-days intensive courses during the first three months of training, with a monthly basis.
  Interventions: Other: Simulation training in Boškoski-Costamagna ERCP Trainer
- Control group (No Intervention): Trainees will undergo routine hands-on clinical ERCP training.

INTERVENTIONS:
Other: Simulation training in Boškoski-Costamagna ERCP Trainer — Coached simulation training in Boškoski-Costamagna ERCP Trainer, by participating in three intensive courses during the first three months of training, with a monthly basis
  Arms: Simulation group

SUMMARY:
The hypothesis of this study is that novice trainees who are offered early simulation training in Boškoski-Costamagna ERCP Trainer in addition to routine hands-on training (intervention group) will demonstrate improved clinical outcomes compared to those undergoing routine hands-on ERCP training only (control group).

DETAILED DESCRIPTION:
Background: Endoscopic retrograde cholangiopancreatography comprises one of the most challenging and complex endoscopic procedures with a steep learning curve. Consequently, adequate training is required to reach competence and perform these procedures safely and with efficacy. To avoid exposing patients to performer-related risk factors, as when trainees practice on real clinical situations, interest in simulator-based endoscopy education is growing. Nonetheless, the validity of simulators is mainly based on endoscopists' subjective opinions about their utility and the implementation of simulators in ERCP training programs is still limited. The Boškoski-Costamagna ERCP Trainer is one of the most appreciated simulation prototypes for ERCP training and has already been demonstrated to have a good face and construct validity. This study aims to evaluate the predictive validity of ERCP Trainer by analyzing the effect of simulation training on the basic ERCP skills of novice ERCP endoscopist trainees and assessing whether it offers an additional benefit to standard training in achieving clinical ERCP competence.

Methods: A prospective, multicenter trial, parallel-arm, randomized controlled trial will be conducted during 1 year. Sixteen "novice" Gastroenterology trainees in high-volume training centers will be randomized into two groups: Group A, intervention group (simulation group with ERCP Trainer) and Group B, control group (no simulation training). Both groups will undergo hands-on clinical ERCP training, supervised by local ERCP trainers, in each trainee's respective Institution. In addition, trainees from Group A will have coached simulation training, by participating in three intensive courses during the first three months of training, with a monthly basis, in Fondazione Policlinico Gemelli, Rome. During the clinical training period, clinical performance evaluation will be systematically evaluated in all ERCPs performed with any degree of trainee involvement. After each trainee completes a minimum of 60 ERCPs, data will be pooled and analyzed. Analysis of overall trainee's competence rates measured by the validated overall trainee's competence rate (TEESAT ERCP score, as primary outcome) and success rate of bile duct cannulation and adverse events rate (secondary outcomes) will be performed.

ELIGIBILITY:
Inclusion Criteria: Gastroenterology trainees from European high-volume training ERCP centers who have previously completed basic endoscopy training but are considered to be novice ERCP endoscopists.

Novice ERCP endoscopists are defined as trainees who have achieved competence in upper gastrointestinal endoscopy, have participated in fewer than 30 ERCPs (with no hands-on experience in ERCP) and are beginning training in a high-volume ERCP center.

Exclusion Criteria: Gastroenterologists with intermediate / advanced expertise in ERCP.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Overall trainee's competence rate | 6 months to 12 months
  The overall trainee's competence rates will be measured by TEESAT ERCP score, graded by supervisor trainer, and the difference between the simulation training group and control group will be compared.

SECONDARY OUTCOMES:
Bile duct cannulation rate | 6 months to 12 months
  Successful biliary cannulation will be specifically defined as deep placement of a guidewire into the common bile duct with contrast visualization.
Adverse events rate | 6 months to 12 months
  Complications include post-ERCP pancreatitis, perforation, bleeding, cholangitis, death and will be assessed up to 72 hours after the procedure, based on symptoms and signs and laboratory tests. Imaging examinations will be performed, if indicated, to rule out complications. Definition of the complications will be assessed on the basis of published criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Teles de Campos, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy